CLINICAL TRIAL: NCT07081555
Title: A First-in-Human Phase 1, Open-label, Two-stage, Randomized Trial to Assess the Safety, Tolerability, and Biodistribution of [177Lu]Lu-ABY-271 in Tumors and Critical Organs in Subjects With HER2-positive Metastatic Breast Cancer
Brief Title: A First-in-Human Phase 1 Safety and Biodistribution of [177Lu]Lu-ABY-271 in Subjects With HER2-positive Metastatic Breast Cancer
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Affibody (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: Affibody AB
Record Dates: First submitted 2025-06-23; First posted 2025-07-23 (Actual); Last update posted 2025-10-01 (Actual); Status verified 2025-06

CONDITIONS: Metastatic Breast Cancer; HER2 + Breast Cancer
Keywords: Radiopharmaceutical; Biodistribution; First-in-human; phase 1; safety
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Intervention Model Description: The trial consists of two parts:
  Part A in which up to 6 subjects will be enrolled sequentially. Part B in which 15 subjects will be randomized to 3 different protein mass dose levels (1:1:1), divided into two sequential cohorts
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Part A (Experimental): [177Lu]Lu-ABY-271
  Interventions: Drug: [177Lu]Lu-ABY-271
- Part B - Cohort 1 (Experimental): [177Lu]Lu-ABY-271 with protein mass dose A
  Interventions: Drug: [177Lu]Lu-ABY-271
- Part B - Cohort 2 (Experimental): [177Lu]Lu-ABY-271 with protein mass dose B
  Interventions: Drug: [177Lu]Lu-ABY-271
- Part B - Cohort 3 (Experimental): [177Lu]Lu-ABY-271 with Protein mass dose C
  Interventions: Drug: [177Lu]Lu-ABY-271

INTERVENTIONS:
Drug: [177Lu]Lu-ABY-271 — A single infusion of [177Lu]Lu-ABY-271

SUMMARY:
This is a FiH phase 1, open-label, two-stage, randomized trial to assess the safety, tolerability, and biodistribution of [177Lu]Lu-ABY-271 in subjects with HER2 positive metastatic breast cancer.

DETAILED DESCRIPTION:
The trial consists of two parts:

Part A in which the uptake of [177Lu]Lu-ABY-271 in tumors and critical organs will be evaluated and up to 6 subjects will be enrolled sequentially.

Part B in which the optimal protein mass dose range (mg) to be utilized in subsequent clinical trials will be evaluated. 15 subjects will be randomized to 3 different protein mass dose levels (1:1:1), divided into two sequential cohorts with different radioactivity levels.

ELIGIBILITY:
Inclusion Criteria:

* Subject has unresectable locally advanced or metastatic breast cancer
* Subject with histologically or cytologically confirmed carcinoma with documented HER2 overexpression (biopsy not older than 2 years): immunohistochemistry (IHC) score 3+; OR 2+ and fluorescence in situ hybridization (ISH) positive
* At least one known tumor lesion ≥ 15 mm
* Eastern Cooperative Oncology Group (ECOG) performance status ≤ 2

Part A only

- Subject is in treatment, or planned to start a new line of standard systemic anti-tumor therapy

Part B only

* Subject has progressive disease, documented radiologically in the last three months
* Subject has received at least 3 lines of standard systemic anti-tumor therapy in the palliative setting
* Subject has received last dose of previous line of systemic anti-tumor therapy, and has no ongoing treatment related toxicities > grade 1 (except alopecia) prior to planned first dose of [177Lu]Lu-ABY-271

Exclusion Criteria:

* Active brain metastases
* Administration of another IMP within 5 half-lives (for experimental biologics: 6 months or 5 half-lives, whichever is longer) of the planned first dose of [177Lu]Lu-ABY-271
* Exposure to any anti-tumor therapy since the last documented progression, including any radiotherapy within 7 days prior to the planned first dose of [177Lu]Lu-ABY-271

Min Age: 18 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 21 (Estimated)
Dates: Start 2025-10-06 (Estimated); Primary Completion 2027-01-01 (Estimated); Study Completion 2028-06-01 (Estimated)

PRIMARY OUTCOMES:
Treatment emergent adverse events | From baseline to the end-of-trial visit, for part A Day 29 and for part B Day 43
Dose Limiting Toxicities | From baseline to the end-of-trial visit, for part A Day 29 and for part B Day 43

SECONDARY OUTCOMES:
Absorbed dose in gray (Gy) per organ and selected tumors | From baseline to day 8
Absorbed dose coefficient (Gy/GBq) per organ and selected tumors | From baseline to day 8
Normalized whole-body effective dose (millisieverts [mSv]/MBq) | From baseline to day 8

CONTACTS AND LOCATIONS:
Locations (3):
- Sweden (3):
  - Sahlgrenska University Hospital, Gothenburg
  - Karolinska University Hospital, Stockholm
  - Akademiska Sjukhuset, Uppsala